CLINICAL TRIAL: NCT04356066
Title: CXCL10 As a Biomarker Of Interstitial Lung Disease in Patients With Rheumatoid Arthritis
Brief Title: CXCL10 As a Biomarker Of ILD in Patients WithRA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Elzahraa Awny Fathy, principle investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: zahraa
Record Dates: First submitted 2020-01-17; First posted 2020-04-22 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-01

CONDITIONS: Interstitial Lung Disease in Patients With Rheumatoid Arthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adult Rheumatoid Arthritis Patient with Interstitial Lung Dise (Other): * History taking: age, sex, disease duration, history of present illness, drug intake, past and family history.
  * Physical examination including thorough clinical examination.
  * Health assessment questionnaire-disability index (HAQ-DI): It is used as a subjective measure of physical function of RA patients (Pincus et al., 1983). There are 20 items in 8 categories: dressing, rising, eating, walking, hygiene, reach, grip, and usual activities (Jessica et al., 2018).
  Interventions: Diagnostic Test: serum cxcl10 by ELISA

INTERVENTIONS:
Diagnostic Test: serum cxcl10 by ELISA — serum sample

SUMMARY:
Rheumatoid arthritis is a chronic inﬂammatory disease that affects the joints, causing symmetric pain, stiffness, swelling, and limited motion and function of multiple joints, its ﬁbro inﬂammatory manifestations may develop in other organs.

DETAILED DESCRIPTION:
Rheumatoid arthritis is complicated by lung manifestations, such as interstitial lung disease which is the most common cause of morbidity and mortality in rheumatoid arthritis patients. Rheumatoid arthritis-interstitial lung disease is a progressive fibrotic disease of the lung parenchyma that includes a broad spectrum of disorders such as nonspeciﬁc interstitial pneumonia, usual interstitial pneumonia , desquamative interstitial pneumonia, cryptogenic organizing pneumonia, diﬀuse alveolar damage, acute interstitial pneumonia, and lymphocytic interstitial pneumonia . Rheumatoid arthritis-interstitial lung disease in which available data indicate that dysregulated inflammatory cascades can elaborate a host of cytokines, chemokines, and growth factors that collectively promote epithelial and endothelial cell damage, angiogenesis, fibroblast differentiation/proliferation, and lung fibrosis . Given the clinical implications of putative signaling cascades involved in these processes, biomarkers that can be used to clarify disease pathogenesis and identify factors governing disease progression are clearly needed .

ELIGIBILITY:
Inclusion Criteria:

1. Adult rheumatoid arthritis patients who fulfilled the 2010 American College of Rheumatology/European league against rheumatism criteria for the classification of Rheumatoid Arthritis.
2. Adult rheumatoid arthritis patients with interstitial lung disease.

Exclusion Criteria:

1. Individuals with other autoimmune diseases (systemic lupus erythematosus, polyarteritis nodosa, dermatomyositis, scleroderma, spondyloarthritis and inflammatory bowel disease).
2. Individuals with hepatitis, Rhinovirus infection, cerebral malaria.
3. Individuals with colorectal carcinoma, syndrome of frailty, vetiligo.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-12-19 (Estimated); Primary Completion 2021-01-19 (Estimated); Study Completion 2022-01-19 (Estimated)

PRIMARY OUTCOMES:
CXCL10 As a Biomarker Of Interstitial Lung Disease in Patients With Rheumatoid Arthritis | 2 years
  serum level

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] 1. Chen J, Doyle TJ, Liu Y, et al. Biomarkers of rheumatoid arthritis-associated interstitial lung disease. Arthritis Rheumatol. 2015;67(1):28-38. doi:10.1002/art.38904 2. Richards TJ, Eggebeen A, Gibson K, et al. Characterization and peripheral blood biomarker assessment of anti-Jo-1 antibody-positive interstitial lung disease. Arthritis Rheum. 2009;60(7):2183-2192. doi:10.1002/art.24631 3. Amigues I, Ramadurai D, Swigris JJ. Current Perspectives On Emerging Biomarkers For Rheumatoid Arthritis-Associated Interstitial Lung Disease. Open Access Rheumatol. 2019;11:229-235. Published 2019 Oct 15. doi:10.2147/OARRR.S166070 4. Vij R, Strek ME. Diagnosis and treatment of connective tissue disease-associated interstitial lung disease. Chest. 2013;143(3):814-824. doi:10.1378/chest.12-0741 5. Castelino FV, Varga J. Interstitial lung disease in connective tissue diseases: evolving concepts of pathogenesis and management. Arthritis Res Ther. 2010;12(4):213. doi:10.1186/ar3097 6. Laragione T, Brenner M, Sherry B, Gulko PS. CXCL10 and its receptor CXCR3 regulate synovial fibroblast invasion in rheumatoid arthritis. Arthritis Rheum. 2011;63(11):3274-3283. doi:10.1002/art.30573 7. Gao B, Lin J, Jiang Z, et al. Upregulation of chemokine CXCL10 enhances chronic pulmonary inflammation in tree shrew collagen-induced arthritis. Sci Rep. 2018;8(1):9993. Published 2018 Jul 3. doi:10.1038/s41598-018-28404-y